CLINICAL TRIAL: NCT05484882
Title: Genomics, Environmental Factors and Social Determinants of Cardiovascular Disease in African Americans Study (GENEFORECAST): Prospective COVID-19 Natural History Study
Brief Title: Genomics, Environmental Factors and Social Determinants of Cardiovascular Disease in African-Americans Study (GENE-FORECAST): Prospective COVID-19 Natural History Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000577; 000577-HG
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-04-16

CONDITIONS: Heart Disease
Keywords: African-American; Cardiovascular Disease; COVID-19; Natural History
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GENEFORECAST: African American men and women residing in the Washington DC area

SUMMARY:
Background:

The COVID-19 pandemic infected and killed African Americans at higher rates than other Americans. Researchers want to understand why.

Objective:

This natural history study will look at how genetic, environmental, and social factors may predict or affect COVID-19 in African Americans. Information from this study will be combined with data from the GENE-FORECAST study.

Eligibility:

African Americans who were previously enrolled in GENE-FORECAST.

Design:

The study includes a telephone interview and 1 visit to the NIH clinic. Participants may engage in either one or both of these activities.

The telephone interview will last 20 minutes. Participants will talk about their experiences during the COVID-19 pandemic.

The clinic visit will last up to 4 hours.

Participants will have a physical exam. They will have blood and urine tests.

They will be tested for COVID-19. A long swab will be inserted into a nostril to get a fluid sample from the back of the nose.

They will have noninvasive tests of their blood vessels. One device used is a pen-like probe placed lightly on the wrist. Another is a rubber sleeve placed around a finger while a blood pressure cuff is used on the arm.

Participants will have a test to measure the electrical activity in their heart. Stickers attached to wires will be placed on their chest, arms, and legs.

Participants will answer more questions about COVID-19. They will talk about their health behavior. They will talk about their family's health and the neighborhood they live in. Other questions will ask how they feel, live, work, and play.

DETAILED DESCRIPTION:
STUDY DESCRIPTION

The objective is to conduct a prospective natural history study of Coronavirus disease 2019 (COVID-19) among a community-based cohort of African Americans enrolled in GENE-FORECAST for whom we have comprehensive psychosocial, clinical, and genetic data collected at baseline. Participants will be invited to take part in a 20-minute computer-assisted telephone interview (CATI) on exposures, attitudes and circumstances during the COVID-19 pandemic and to undergo a clinic visit for a physical exam, vascular function tests and biospecimen collection. We will identify social, clinical and genetic risk factors for COVID-19 and examine the interplay between social determinants of health and personal risk profiles to better understand the disparate burden of COVID-19 in the African American community. It is hypothesized that exposure to the SARS-CoV-2 virus and the development of COVID-19 will be associated with social and neighborhood factors, and that SARS-CoV-2 infection will adversely affect vascular function.

OBJECTIVES

Primary Objectives:

1. Define the effect of social factors (e.g., socio-economic status; neighborhood characteristics) on exposure to SARS-CoV-2 and the development of COVID-19.
2. Define the effect of SARS-CoV-2 infection and the development of COVID-19 on vascular function (e.g., pulse wave velocity).
3. Examine how social factors influence the effect of SARS-CoV-2 and COVID-19 on vascular function.

Secondary Objectives:

1. Examine the effects of SARS-CoV-2 infection and COVID-19 on epigenome (whole-blood), transcriptome, (whole-blood, plasma

   microvesicles, urine), peripheral blood mononuclear cell (PBMC) single-cell RNA-seq, biomarker profile (e.g., CRP; d-dimer), cardiac function (EKG) and leukocyte telomere length.
2. Examine how social factors influence the effect of SARS-CoV-2 infection and COVID-19 on transcriptome and epigenome.

ENDPOINTS

Primary Endpoints:

SARS-CoV-2 infection

Vascular function (e.g., pulse wave velocity; vascular stiffness indices; reactive hyperemia)

Secondary Endpoints:

Transcriptome (whole-blood, plasma microvesicles, urine)

Epigenome (whole-blood)

PBMC single-cell RNA-seq

Leukocyte telomere length

Electrocardiogram (EKG)

Biomarker profile (CRP, D-Dimer, ACE-2, HS-Troponin)

ELIGIBILITY:
* INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Self-identified African American men and women who previously enrolled in GENE-FORECAST, completed baseline activities and gave permission for recontact through the GENE-FORECAST protocol.
* Stated willingness to participate in study procedures.
* Ability of subject to understand and the willingness to give verbal informed consent for the CATI and the ability to understand and the willingness to sign a written informed consent document for the clinic visit.

Individuals eligible for this protocol are previous GENE-FORECAST participants, all of whom are English speakers. Therefore, by default, this study includes only English speakers.

EXCLUSION CRITERIA

Only individuals who completed the baseline protocol of GENE-FORECAST and gave permission for recontact through the GENE-FORECAST protocol will be invited to participate. Among this group, there are no exclusions for this study except those who are pregnant.

Ages: 21 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 650 African American men and women residing in the metropolitan DC area who previously competed baseline activities in the GENE-FORECAST protocol. Participants will be at least 21 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Define the effect of SARS-CoV-2 infection and the development of COVID-19 on vascular function (e.g., pulse wave velocity). | 48 month
  Vascular function (e.g., pulse wave velocity; vascular stiffness indices; reactive hyperemia)
Examine how social factors influence the effect of SARS-CoV-2 and COVID-19 on vascular function. | 48 month
  African Americans are disproportionately affected by SARS-CoV-2 infection and COVID-19. There are well-documented socioeconomic inequalities that contribute to this increased vulnerability. The disparate burden of disease demands a multidimensional approach informed by social determinants of health, geography (neighborhood), and personalized risk profiles. Among the social, environmental, clinical and genetic factors likely to be important for COVID-19 risks and outcomes, there is little understanding of the relative importance of these factors among African Americans and how they interact to affect morbidity and mortality.
Define the effect of social factors (e.g., socio-economic status; neighborhood characteristics) on exposure to SARS-CoV-2 and the development of COVID-19 | 48 month
  Vascular function (e.g., pulse wave velocity; vascular stiffness indices; reactive hyperemia)

SECONDARY OUTCOMES:
Examine how social factors influence the effect of SARS-CoV-2 infection and COVID-19 on transcriptome and epigenome. | 48 month
  Biomarker profile (CRP, D-Dimer, ACE-2, HS-Troponin) * Analyses of all of the above endpoints will use change in values from baseline GENE-FORECAST to current measures.
Examine the effects of SARS-CoV-2 infection and COVID-19 on epigenome (whole-blood), transcriptome, (whole-blood, plasma microvesicles, urine), peripheral blood mononuclear cell (PBMC) single-cell RNA-seq, biomarker profile (e.g., CRP; d-dimer),... | 48 month
  Transcriptome (whole-blood, plasma microvesicles, urine) Epigenome (whole-blood) PBMC single-cell RNA-seq Leukocyte telomere length

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Westat, Inc., Rockville, Maryland

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000577-HG.html